CLINICAL TRIAL: NCT06348654
Title: Application of a New Digital Person-based Care (PbC) Model for the Treatment of Patients With HER2-negative Advanced Breast Cancer
Brief Title: New Digital Person-based Care Model in Patients With HER2-negative Advanced Breast Cancer
Acronym: InPERSON
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FABI ALESSANDRA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6392
Record Dates: First submitted 2024-03-20; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Narrative Medicine; HER2-negative Breast Cancer; Patient Satisfaction
MeSH Terms: conditions — Breast Neoplasms; Narrative Medicine; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: introduction of digital listening may improve the quality of life of patients withe breast cancer — Introduction of a digital listening and communication pathway aimed at improving the quality of life of patients with advanced HER2-negative breast cancer

SUMMARY:
The goal of the InPerson study is to employ all resources in a digital listening platform to benefit the quality of life of patients (QoL) with advanced HER2-negative breast cancer.

The care pathway of patients with this type of disease represents an optimal setting for the implementation of an innovative narrative medicine pathway that, aided by integrative therapies, aims to support and accompain them in their treatment journey with a continuum of care. Moreover, the narrative medicine platform will implement the actual "static" way to define QoL with the classic Patient-Reported Outcomes (PROs) questionnaires, that reflect the patient status at a certain time point and not as a dinamic entity. It is on the basis of these assumptions that the present application project on the use of the DNMLAB digital narrative diary in the oncology department of the Fondazione Policlinico Gemelli was born.

DETAILED DESCRIPTION:
In recent years, the health care system has undergone significant changes that have led to the emergence of a person-centered medicine paradigm. In this new scenario, outcomes of care pathways are evaluated not only on the basis of clinical outcomes but also in terms of the impact on patients' quality of life. Due to therapeutic advances, it therefore becomes increasingly necessary to adopt integrated, empathic and person-centered clinical approaches that also take into account patients' needs and expectations for care.

New measurement tools that assess also the patient's perspective have been introduced into clinical practice.

Among these new tools are Patient-Reported Outcome Measures (PROMs), aimed at determining patients' perceived quality of life during treatment and follow-up. Systematic collection of patient-reported outcomes has indeed been proven to be a valid, reliable, and accurate methodology in oncology, both for assessing treatment outcomes and monitoring drug toxicity, and for avoiding all those cases where impacts and symptoms are overlooked or underestimated by clinicians.

However, currently approved and standardized questionnaires do not comprehensively inform clinicians about how the disease and treatments affect the patient's care pathway.

In this context, narrative medicine, on the other hand, has proven to be a valid and reliable methodology capable of integrating the patient's perspective into standard clinical assessment.

Qualitative narrative medicine methodologies have been recognized as useful and effective to the extent that they allow clinicians to access the existential and emotional components of patients' experience of care, and for their ability to enrich the information expressed in standardized questionnaires. Narrative methodologies thus make it possible to capture perceptions of quality of life, and thus to capture a highly subjective dimension influenced by each individual's needs and expectations (e.g., relative deprivation).

Narrative medicine has also been shown to be feasible and reliable in improving doctor-patient communication and promoting bio-psycho-social personalization of the care pathway, particularly when used in combination with digital listening tools, such as the digital narrative diary. Studies on digital narrative medicine in oncology have shown the potential of digital platforms in promoting listening to patient needs, especially when listening is done by a multidisciplinary care team throughout the care pathway. It has also been seen how digital has a positive impact not only on the patient but also, more broadly, on the entire care team.

The transition from a traditional, disease-centered model of care to a new, more person-centered model of care has since led to the introduction of integrative medicine in cancer treatment centers. Through the rational and evidence-based use of lifestyle, psychological support, and complementary therapies, integrative medicine promotes better control of side effects, greater adherence to treatment protocols, and optimization of patients' quality of life throughout the care pathway. In the case of breast cancer, integrative oncology combines conventional cancer treatments with integrative therapies in order to support women in their bio-psycho-social dimensions, thus providing effective and minimally invasive responses to complex and sometimes unmet health needs.

ELIGIBILITY:
Inclusion Criteria:

* HER2-negative advanced disease undergoing first- or second-line oncological treatment combined with integrative therapies;
* Age ≥18 years;
* Knowledge of Italian language;
* Life expectancy ≥24 weeks.

In case the patient is unable to actively participate, the caregiver can act as a vicarious narrator and contribute to the study by supplementing the patient's contribution.

Exclusion Criteria:

* ECOG Performance Status >2;
* Inability to participate in the study due to psychiatric disorders;
* Unavailability of an e-mail account or unwillingness to use web-based tools.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population refers to women with HER2-negative advanced breast cancer (IHC score 0, 1+ or 2+ with unamplified FISH/SISH) in first- or second-line treatment, with advanced disease, undergoing cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Standardized quality-of-life measurement | 12 months
  The integration of standardized quality-of-life measurement with the patient's subjective narrative through the application of validated narrative medicine methodologies.
  Primarily QoL questionnaires from EORTC QLQC-30 and QLQ-BR23, implemented with digital narrative tehniques.
Perceived quality of life | 12 months
  The improvement of the perceived quality of life of patients with advanced breast cancer,Primarily QoL questionnaires from EORTC QLQC-30 and QLQ-BR23, implemented with digital narrative tehniques.
Personalization of the care pathway | 12 months
  Personalization of the care pathway through integrative therapies, based on patients' needs, attitudes and lifestyles. This does not necessarily need standardized questionnaires, because if the patient raise concern about a sign or symptom, this will be properly evaluated with the last CTCAE available version.
Quality of the patient-physician relationship. | 12 Months
  The improvement of the quality of the patient-physician relationship. This is not necessary linked to a standardized evaluation method or solely to an improvement in QoL measured with the already cited questionnaires. Dedicated perception scales will be created by the digital narrative team to explore if the proposed methods are feasible.

SECONDARY OUTCOMES:
Interaction between multidisciplinary teams | 12 months
  The strengthening of interaction between multidisciplinary teams. Personalization of the care pathway implicitly needs the involvement of other professional figures: psychologist, antropologist, radiotherapist, dietician, integrative care specialist. Based on this, the team will try to develop a "holistic" care pathway, tailored on the single patient.
Patient involvement and compliance in the care pathway | 12 Months
  The validation of digital tools to introduce innovative models of patient involvement and compliance in the care pathway. The continuos feedback from the oncologist based on the narrative diary will help the clinician to estimate the treatment compliance and the possible side effects.
lifestyles best suited to positively affect quality of life | 12 Months
  The enhancement of communication processes aimed at informing metastatic patients about lifestyles best suited to positively affect quality of life. Through the collaboration with the integrative care team, if needed, a change in lifestyle with a structured schedule will be proposed to each single patient.
Awareness of disease condition | 12 Months
  Increasing patients' awareness of their disease condition, the effects of treatment, and the care needs that may arise during treatment. The diary gives to the patient the opportunity to develop an introspective dimension of the disease, and stimulates her to properly elaborate the steps of the care pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Fabi Alessandra, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Roma